CLINICAL TRIAL: NCT02464189
Title: Assessment of Asthma Knowledge Perception in Parents of Asthmatic Children. Pilot Study by Means of Q-KAP ( Questionnaire on Knowledge, Attitudes and Practices )
Acronym: Q-KAP
Status: Completed | Type: Observational
Sponsor: Stefania La Grutta, MD (Other)
Responsible Party: Sponsor-Investigator, Stefania La Grutta, MD, Stefania La Grutta, MD. Senior Researcher. Coordinator of Pediatric Allergy and Asthma Research Group. Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Organization: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Other Study IDs: 10/2014
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with asthma
  Interventions: Other: Q-Kap

INTERVENTIONS:
Other: Q-Kap

SUMMARY:
The aim of this study is to assess the knowledge, the attitudes and the practices of parents of asthmatic children.

DETAILED DESCRIPTION:
The aim of this study is to assess the knowledge, the attitudes and the practices of parents of asthmatic children.

The study proposes the validation of Q- KAP by means of the recruiting of 390 parents of asthmatic children, recruited in the outpatient clinic of Pediatric Allergology & Pulmonology (PAP) of Respiratory Disease Research Center (RDRC) within the Institute of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (RDRC-IBIM CNR), Italy.

Q-KAP will be given to one of the parents during their children medical examination. Q-KAP is a multiple answer questionnaire investigating on knowledge, attitudes and practices for what concerns Asthma.

At the end of the recruitment time, data will be stored and analyzed in a dataset.

The expected result is the identification of a tool able to assess knowledge, attitudes and practices of asthmatic children parents, but also the identification of a tool able to identify two groups of parents (well-experienced and bad-experienced) to assess if there is a link between a low degree of knowledge and a bad control of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Asthma

Exclusion Criteria:

* No consent by parents

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 390 asthmatic children, recruited in the outpatient clinic of Pediatric Allergology & Pulmonology (PAP) of Respiratory Disease Research Center (RDRC) within the Institute of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (RDRC-IBIM CNR), Italy.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2015-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Knowledge, attitudes and practices of parents of asthmatic children assessment. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Biomedicine and Molecular Immunology, IBIM, Palermo, Italy

IPD SHARING:
Plan to Share IPD: Yes
The IPD collected will be available on December 2016.
  The following participant data will be shared:
  * Asthma severity level
  * Asthma control level
  * Pulmonary function tests
  * Demographic characteristics All IPD will be obtained from statistical analysis on the dedicated database in which all data are stored.